CLINICAL TRIAL: NCT02537158
Title: Sorafenib and TACE as Adjuvant Therapy for MVI in HCC Patients After Radical Resection:a Non-randomized Controlled Trial
Brief Title: Sorafenib and TACE as Adjuvant Therapy for MVI in HCC Patients After Radical Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xinyu Bi, Xinyu Bi, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-077
Record Dates: First submitted 2015-08-29; First posted 2015-09-01 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: sorafenib; transcatheter arterial chemoembolization; hepatocellular carcinoma; microvascular invasion
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sorafenib group (Experimental): sorafenib group patients will accept sorafenib therapy for one year（400 mg bid,orally).
  Interventions: Drug: Sorafenib
- TACE group (Experimental): TACE group patients will accept TACE therapy once at a month after resection.
  Interventions: Procedure: TACE
- control group (No Intervention): Control group patients will not accept any intervention,except necessary supportive treatment.

INTERVENTIONS:
Drug: Sorafenib — sorafenib group patients will accept sorafenib therapy for one year（400 mg bid,orally).
  Arms: sorafenib group
Procedure: TACE — TACE group patients will accept TACE therapy once at a month after resection.
  Arms: TACE group

SUMMARY:
This study is a prospective non-randomized controlled study. The purpose of this study is to evaluate the validity and safety of sorafenib and transcatheter arterial chemoembolization (TACE) for microvascular invasion (MVI) in hepatocellular carcinoma (HCC) patients after radical surgery.

DETAILED DESCRIPTION:
HCC is the sixth most common malignancy worldwide.Selected patients with HCC are candidates for potentially curative therapy, such as hepatic resection and liver transplantation. Nevertheless,tumor recurrence is 70 % at 5 years after resection and 15-30 % after liver transplantation,leading to tumor-related death.MVI is currently one of the most critical factors predictive of HCC recurrence.There are no approved effective interventional measures to improve the outcome of this patients with MVI.The purpose of this study is to explore the validity and safety of sorafenib and TACE for MVI in HCC patients after radical resection.The candidates will be assigned to sorafenib group (about 30 cases),TACE group (about 30 patients) and control group (about 30 cases)，according to the willingness of the subject.All patients will be followed up for 3 years and Recurrence-free survival and overall survival will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age;
* The liver tumor has been radically resected;
* Postoperative pathology proved to be hepatocellular carcinoma with negative margin and microvascular invasion;
* Imaging evaluations(CT/MRI) were performed at 1 month after the resection and no area of enhancement was seen;
* Child-Pugh A;
* Eastern Cooperative Oncology Group(ECOG) body condition score (PS) 0-1;
* Then patients understand and voluntarily signed a written informed consent;

Exclusion Criteria:

* Recurrent HCC;
* pathology-proved multifocal HCC or HCC with satellite nodules;
* Tumor thrombus in portal vein or inferior vena cava trunk;
* Patients with extrahepatic metastasis found by radiologic or pathologic examination;
* severe dysfunction of the heart, kidney, or other organs.The patients cannot tolerate TACE or sorafenib after general assessment of the situation;
* Enrolled in other clinical study at the same time;
* Previously treated with other antitumor treatments except the resection;
* The researchers believe that the patient does not fit this study;
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival | 36 month

SECONDARY OUTCOMES:
overall survival | 36 month

CONTACTS AND LOCATIONS:
Overall Officials: Xinyu Bi, Doctor, Study Director — Cancer Hospital and Institute, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital and Institute, Chinese Academy of Medical Sciences, Beijing, China

REFERENCES:
- [Background] Rodriguez-Peralvarez M, Luong TV, Andreana L, Meyer T, Dhillon AP, Burroughs AK. A systematic review of microvascular invasion in hepatocellular carcinoma: diagnostic and prognostic variability. Ann Surg Oncol. 2013 Jan;20(1):325-39. doi: 10.1245/s10434-012-2513-1. Epub 2012 Nov 13. PMID 23149850
- [Background] Sumie S, Nakashima O, Okuda K, Kuromatsu R, Kawaguchi A, Nakano M, Satani M, Yamada S, Okamura S, Hori M, Kakuma T, Torimura T, Sata M. The significance of classifying microvascular invasion in patients with hepatocellular carcinoma. Ann Surg Oncol. 2014 Mar;21(3):1002-9. doi: 10.1245/s10434-013-3376-9. Epub 2013 Nov 20. PMID 24254204
- [Background] Roayaie S, Blume IN, Thung SN, Guido M, Fiel MI, Hiotis S, Labow DM, Llovet JM, Schwartz ME. A system of classifying microvascular invasion to predict outcome after resection in patients with hepatocellular carcinoma. Gastroenterology. 2009 Sep;137(3):850-5. doi: 10.1053/j.gastro.2009.06.003. Epub 2009 Jun 12. PMID 19524573
- [Background] Zhu YB, Xu X, Zheng SS. [Association of microvascular invasion with recurrence and prognosis of patients with small hepatocellular carcinoma undergoing liver transplantation]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2014 Nov;43(6):658-63. doi: 10.3785/j.issn.1008-9292.2014.11.004. Chinese. PMID 25644564
- [Background] Shirabe K, Toshima T, Kimura K, Yamashita Y, Ikeda T, Ikegami T, Yoshizumi T, Abe K, Aishima S, Maehara Y. New scoring system for prediction of microvascular invasion in patients with hepatocellular carcinoma. Liver Int. 2014 Jul;34(6):937-41. doi: 10.1111/liv.12459. Epub 2014 Jan 24. PMID 24393295
- [Background] Meniconi RL, Komatsu S, Perdigao F, Boelle PY, Soubrane O, Scatton O. Recurrent hepatocellular carcinoma: a Western strategy that emphasizes the impact of pathologic profile of the first resection. Surgery. 2015 Mar;157(3):454-62. doi: 10.1016/j.surg.2014.10.011. Epub 2014 Nov 6. PMID 25633732